CLINICAL TRIAL: NCT02927353
Title: A Phase 1 Pharmacokinetic Bioequivalence Study of DMB-3113 and Adalimumab in Healthy Japanese Adult Male Subjects
Acronym: DMB-3113-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Meiji Seika Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DMB-3113-1
Record Dates: First submitted 2016-10-05; First posted 2016-10-07 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2016-06

CONDITIONS: Healthy Volunteer
Keywords: Bioequivalence, Biosimilarity, Pharmacokinetics, adalimumab
MeSH Terms: interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DMB-3113 (Experimental): adalimumab biosimilar
  Interventions: Drug: DMB-3113
- adalimumab (Active Comparator): adalimumab
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: DMB-3113 — subcutaneously injected in a single dose of 40 mg.
  Arms: DMB-3113
Drug: Adalimumab — subcutaneously injected in a single dose of 40 mg.
  Arms: adalimumab

SUMMARY:
To determine the pharmacokinetic bioequivalence of DMB-3113 and adalimumab and to confirm the safety of the study drug in healthy Japanese adult male subjects

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Japanese male adults;
2. The Body Mass Index (BMI) of the subjects must be from 17.6 to 26.4 kg/m2 at the time of the screening test;and
3. Subjects must take a screening test within the 4 weeks before the date of administration of the study drug; subjects must take a screening test before the date of administration of the study drug and exhibit no clinically abnormal findings in the judgment of the investigator or any of the subinvestigators

Exclusion Criteria:

1. Concurrent or history of potentially fatal infections such as opportunistic infections, including sepsis, pneumonia, and fungal infection;
2. Individuals with history of tuberculosis or diagnosed with tuberculosis by interview, chest X-ray examination, or interferon-gamma release assay;
3. Concurrent or history of demyelinating disease (multiple sclerosis, etc.);
4. Concurrent or history of congestive cardiac failure;
5. Concurrent or history of allergic symptoms such as asthma bronchial, drug-induced rash, and urticaria, which, in the judgment of the investigator or any of the subinvestigators, may affect participation in this clinical study; or
6. Concurrent or history of cardiac, hepatic, renal, gastrointestinal, respiratory, and/or hematological function disorders, which, in the judgment of the investigator or any of the subinvestigators, may affect participation in this clinical study

Ages: 20 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2016-08; Primary Completion 2017-01-17 (Actual); Study Completion 2017-01-17 (Actual)

PRIMARY OUTCOMES:
Area under the serum concentration-time curve (AUC) from 0 to final sampling time point | Day 1 to Day 71
AUC from 0 to infinity | Day 1 to Day 71
Maximum serum concentration (Cmax) | Day 1 to Day 71

SECONDARY OUTCOMES:
AUC from 0 to the last measurable concentration | Day 1 to Day 71
Time to reach the peak concentration (tmax) | Day 1 to Day 71
Mean residence time (MRT) from 0 to final sampling time point | Day 1 to Day 71
MRT from 0 to infinity | Day 1 to Day 71
Elimination rate constant (kel) | Day 1 to Day 71
Elimination half life (t1/2) | Day 1 to Day 71
Observed clearance (CL/F) | Day 1 to Day 71
Observed volume of distribution (V/F) | Day 1 to Day 71
Incidence of adverse events | Day 1 to Day 71

CONTACTS AND LOCATIONS:
Overall Officials: Hideki Fushimi, Manager, Study Director — Meiji Seika Pharma Co., Ltd.
Locations (1):
- Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: No